CLINICAL TRIAL: NCT03922984
Title: A Prospective Study to Evaluate Quantitative Non-Contrast Perfusion Using Arterial Spin Labeled Magnetic Resonance (MR) Imaging for Assessment of Therapy Response in Glioblastoma
Brief Title: Non-Contrast Perfusion Using Arterial Spin Labeled MR Imaging for Assessment of Therapy Response in Glioblastoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ananth Madhuranthakam, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU 032018-079; 1U01CA207091-01A1 (NIH)
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Glioblastoma
Keywords: magnetic resonance imaging, arterial spin labeling
MeSH Terms: conditions — Glioblastoma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glioblastoma Patients (Experimental): Patients with histologically proven glioblastoma will undergo enhanced MRI with arterial spin labeling at weeks 0, 3, 6, 10, 18, 26, and 34 after beginning standard of care treatment.
  Interventions: Procedure: MRI with Arterial Spin Labeling (ASL)

INTERVENTIONS:
Procedure: MRI with Arterial Spin Labeling (ASL) — Week 0 (Before initiation of chemoradiation): MRI with ASL will be performed along with patient's standard of care imaging session Week 3: contrast-enhanced research MRI with ASL Week 6: contrast-enhanced research MRI with ASL Week 10: MRI with ASL will be performed along with patient's standard of care imaging session Week 18: MRI with ASL will be performed along with patient's standard of care imaging session Week 26: MRI with ASL will be performed along with patient's standard of care imaging session Week 34: MRI with ASL will be performed along with patient's standard of care imaging session

SUMMARY:
MRI including ASL will be performed before, during and after the treatment, in a total of 7 MRI sessions until 8 months after the first session. Thereafter, patients will be followed through standard clinical examinations for the next 3 years or until demise, whichever occurs first.

Clinically, GBM patients are imaged every 8-weeks, beginning at 10 weeks after the completion of chemoradiation, since morphological (i.e. size) changes are not anticipated earlier. However, our preliminary experience and others have shown functional changes including perfusion and diffusion as early as 3-weeks after the initiation of the treatment . Thus, our T10, T18, T26 and T34 MRI sessions will be performed along with the clinical imaging sessions, while the T3 and T6 MRI sessions will be performed additionally for this proposal. All MR imaging sessions will be scheduled within ±1 or ±2 weeks of the target time period, as indicated in the table.

MRI including ASL will be performed before, during and after the treatment, in a total of 7 MRI sessions until 8 months after the first session. The research MR imaging may take approximately an additional 15 minutes per each imaging session. However, the T3, and T6 MR imaging sessions will be performed additionally for the purpose of this study, with each taking approximately one hour. Thereafter, patients will be followed through standard clinical examinations for the next 3 years or until demise, whichever occurs first.

DETAILED DESCRIPTION:
Glioblastoma (GBM) represents about 15% of all primary brain tumors with approximately 19,000 new cases diagnosed annually. The one-, five- and ten-year survival rates for patients with GBM is 37.2%, 5.1% and 2.6% from diagnosis respectively, making it one of the most lethal cancers known, among all cancers. GBMs can be challenging to treat and new cancer therapies are continuously being developed for GBM treatment.

The high cost and potential risks associated with human trials for these experimental therapies have emphasized the need for sensitive monitoring of tumor response. Imaging approaches can play an important role in the evaluation and selection of potential new therapies with non-invasive longitudinal monitoring of treatment response. Currently, the radiological assessment of treatment outcomes predominantly relies on morphological (i.e. size) changes using the Response Evaluation Criteria in Solid Tumors (RECIST) and other similar scores. This is a major limiting factor as the effects of many therapeutic agents at the microscopic level precede the eventual changes in tumor size. One such tumor property that has gained increased attention is angiogenesis, which has been shown to support tumor proliferation and infiltration. Increasing numbers of clinical trials have begun targeting tumor vascular supplies either directly inhibiting angiogenesis (e.g. antiangiogenic therapy) or indirectly disrupting cell proliferation and eventually angiogenesis (e.g. cytotoxic chemoradiation). Such clinical trials and the eventual clinical use of these therapies would be greatly assisted by the availability of robust imaging indicators of angiogenesis (i.e. tissue perfusion).

Positron Emission Tomography (PET) using 15O-labeled water (15O-PET) is considered the gold standard for non-invasive measurement of tissue perfusion. However, the use of 15O-PET requires a cyclotron in close proximity to PET to produce short lived 15O-water (half life 2.4 min), limiting its applicability in clinical settings. Alternative imaging techniques include ultrasound using microbubbles, perfusion computed tomography (CT) using iodinated contrast agent and perfusion MRI using gadolinium based contrast agents. All of these techniques require exogenous agents, restricting their use in longitudinal monitoring of treatment response.

Arterial spin labeled (ASL) MRI has recently emerged as a quantitative imaging (QI) method to measure perfusion (or capillary blood flow) without the administration of exogenous contrast agents. ASL magnetically "labels" the highly permeable water in the blood as a tracer and measures their accumulation in the tissue of interest, without injecting any exogenous contrast. Various versions of ASL have been validated in animals using microspheres, and in humans using 15O-PET in the brain. ASL also has a number of advantages compared to dynamic contrast enhanced (DCE) and dynamic susceptibility contrast (DSC) based MR perfusion measurements. Specifically, ASL does not require exogenous agent alleviating the concerns of gadolinium accumulation or nephrogenic systemic fibrosis (NSF) in patients with impaired renal function and, unlike DCE/DSC, the contribution of vascular permeability to ASL measured perfusion is negligible enabling absolute perfusion quantification in physiological units (ml/100g/min).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven GBM
* Newly diagnosed GBM. Prior surgery is allowed, but should not have started any other treatment such as chemotherapy, radiation treatment, and anti-angiogenic therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Women of child-bearing potential must agree to undergo a urine pregnancy screening per standard Radiology departmental protocol, in place to prevent imaging of pregnant patients. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: 1) Has not undergone a hysterectomy or bilateral oophorectomy; or 2) Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Scheduled to undergo chemoradiation.

Exclusion Criteria:

* Subjects who have had prior chemotherapy or radiotherapy.
* Subjects may not be receiving any other investigational agents at the time of enrollment.
* Subjects must not be pregnant since pregnancy is a contraindication to administration of gadolinium-based contrast agents.
* Any contraindication to MRI per Radiology Department's routine protocol, e.g. MRI-incompatible objects, including but not limited to medical devices (e.g. pacemakers, automated implantable cardioverter defibrillators, etc.) and other foreign bodies.
* Known severe allergic reaction to Gadolinium-based contrast agents.
* Patients with sickle cell disease and patients with other hemolytic anemias (low red blood count in body).
* Patients with uncontrollable claustrophobia, severe lower back pain, and uncontrollable tremors, to the point that it would render them unable to tolerate an MRI study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Change in perfusion within enhancing tumor | Baseline to 3 weeks
  Will determine changes in ASL measured tumor perfusion is associated with treatment response, measured as time to progression. One-sample correlation test will be used to determine the correlation between change in ASL measured tumor perfusion (baseline to 3 weeks) and time to progression. The correlations will be measured and compared using Pearson's correlation coefficient along with 95% confidence interval.
Progression Free Survival (PFS) | Up to 3 years
  Will determine if changes in ASL measured perfusion is associated with PFS. PFS will be correlated with baseline perfusion and post-treatment changes at 3-, 6- and 10-weeks compared to baseline using univariable and multivariable Cox regression models. Will determine whether changes in ASL measured tumor perfusion as a continuous variable within enhancing tumor from baseline to 3-, 6-, and 10-weeks after initiation of chemoradiation is associated with PFS. The hazard ratio and its 95% confidence interval will be presented.

SECONDARY OUTCOMES:
ASL measured perfusion within enhancing tumor | Baseline
  Will determine if ASL measured tumor perfusion at baseline is associated with treatment response, measured as time to progression. One-sample correlation test will be used to determine the correlation between baseline ASL measured tumor perfusion and time to progression. The correlations will be measured and compared using Pearson's correlation coefficient along with 95% confidence interval.
Overall Survival (OS) | Up to 3 years
  Will determine if changes in ASL measured perfusion is associated with OS. OS will be correlated with baseline perfusion and post-treatment changes at 3-, 6- and 10-weeks compared to baseline using univariable and multivariable Cox regression models. Will determine whether changes in ASL measured tumor perfusion as a continuous variable within enhancing tumor from baseline to 3-, 6-, and 10-weeks after initiation of chemoradiation is associated with OS. The hazard ratio and its 95% confidence interval will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Ananth Madhuranthakam, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No